Official Title: Effect of Emotion Mindsets on Emotion Processing: A Multilevel Experimental

Investigation

NCT Number: 03978871

Date of final version of consent: July 29th, 2020

# UNIVERSITY OF ILLINOIS AT URBANA-CHAMPAIGN



#### PARENT CONSENT FORM

**Title of study:** Study of Teen Emotion Processing (STEP)

Principal Investigator/s: Dr. Karen Rudolph, Dr. Wendy Heller, & Dr. Sepideh Sadaghiani

Contact information is listed on p. 3.

**Department/s:** Psychology, University of Illinois at Urbana-Champaign

## **Research project:**

The purpose of this research is to examine emotion processing in adolescents and to help individuals develop adaptive ways of dealing their emotions. The study involves completing questionnaires, viewing video clips, and participating in a debriefing discussion with a staff member. Study participation will take approximately 150 minutes.

### **Procedures:**

- 1) You will be asked to fill out a few surveys, including demographic information and measures about emotions. Completing the surveys will take about 10-15 minutes. You may review all of your child's measures prior to her participation.
- 2) Your child will be asked to fill out a number of questionnaires. The types of topics addressed in the questionnaires include emotions, behaviors, and experiences, including questions specific to her experiences during the COVID-19 pandemic. Example questions include "I felt unhappy or miserable," "I cheer up quickly," and "How many people close to you were diagnosed with COVID." These questions should take no more than 30 minutes to complete. The questionnaires can be completed using a secure on-line website or on paper.
- 3) Your child will be asked to participate in a role play where they will talk about friendships. During this task, your child will be asked to make a four-minute speech in front of research staff while facing a camera. This portion of the study will be recorded via video. This recording will be kept completely secure and will only be shared with researchers on our team for research purposes. While the completion of this task has the potential to cause mild discomfort, it is expected to be similar to any act of public speaking. We will check in with your child at the end of the visit, and if feelings of discomfort persist we will follow-up with you and her the following day.
- 4) Your child will be asked to view brief video clips and rate how they feel after viewing them. Some of the video clips she will view are moderately negative. While viewing these video clips may cause mild discomfort, they do not pose any risk. The images your child views may cause mild discomfort because they may remind your child of negative experiences in her own life. If your child reports higher than baseline ratings on a measure of her emotions at the end of the study, we will follow-up with you and her the following day.

- 5) Your child will complete a computer task in which she pushes a button whenever she sees a letter except the letter "x."
- 6) Your child will be asked to complete a computer-administered session in which she will learn about adolescent development and some basic information about the brain. We will also ask your child to provide information to younger adolescents based on what she learned. This computer session will last approximately 30 minutes.
- 7) Finally, project staff will conduct a debriefing session with your child. The purpose of this session is for our staff to ask questions and receive feedback from participants on certain measures and aspects of our study. For example, project staff may ask if any words or items were confusing to your child. Project staff may take hand-written notes of her responses during this part.

All procedures will be employed with sensitivity to your child's feelings. To avoid any discomfort, your child may skip questions she does not want to answer. Her participation in this study is voluntary, and she may withdraw from the study at any time without penalty.

Your child will be offered breaks periodically throughout the study session. She is encouraged to notify the researchers that she needs to take a break at any time. Restrooms and drinking water will be available during study sessions.

#### **Remuneration:**

Your child will receive \$50 for her participation. If your child's participation is discontinued (by you, your child, or the experimenter), your child will be paid according to her level of participation. You will not receive remuneration for your participation as you will complete a small subset of measures.

#### **Risks & Benefits:**

Your child will be asked to report on sensitive topics, including their emotions. While these questions are sensitive in nature, answering them does not pose any expected risk to your child. Your child's responses will be completely confidential and voluntary and your child may choose not to respond to any questions that she is uncomfortable with. The answers to your child's questions will not be shared with anyone except our research team unless we are concerned about your child's or someone else's safety.

There is no direct personal benefit to participating in this study. However, your child's participation provides the investigator with a greater understanding about emotional development in youth. The study results may be used to help other people in the future.

# **Confidentiality:**

All possible steps have been taken to assure your child's privacy. The experimenter will assign your child an arbitrary code number which will be used throughout the study. Only this code (and never your child's name) will be used when analyzing or reporting the data. Any identifying information will be kept in a locked location in the Investigator's laboratory. In addition, laws and University rules might require that the research data be made available to the following groups: 1) representatives of the University committee and office that reviews and approves research studies, such as the Institutional Review Board (IRB) or Office for Protection of Research Subjects; 2) representatives of the state and University responsible for ethical, regulatory, or financial oversight of research; and, 3) research collaborators at the Biomedical Imaging Center. Anyone who accesses the research data will be required to maintain the confidentiality of any and all participants.

# Voluntary participation and withdrawal:

Participation in the research is voluntary. Your child is free to stop participating at any time. If your child

#### A1. Parent Consent

chooses not to volunteer, or if the research is ended for any reason by you, your child, or the researchers, it will have no effect on any other benefits to which your child is entitled. If your child is a student at the University of Illinois, her decision to participate, decline, or withdraw from participation will have no effect on her grades at, status at, or future relationships with the university.

# **Dissemination of findings:**

The results of the research may be published, and presented at lectures and professional meetings, but your child will not be identified in any such publication or presentation.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify your child. At most, the Web site will include a summary of the results of the research project. You can search this website at any time.

#### **Contact Information:**

You will be given a copy of this consent form for your records. If at any time, either now or later, you have a question, please feel free to ask it. If you have questions or concerns regarding your child's rights as a participant in this study, please contact the University of Illinois Institutional Review Board office at (217) 333-2670 or <a href="mailto:irb@illinois.edu">irb@illinois.edu</a>. If you have any questions about this particular study, you may contact Dr. Karen Rudolph at (217)333-8624 or <a href="mailto:krudolph@illinois.edu">krudolph@illinois.edu</a>, Dr. Wendy Heller at (217)244-8249 or <a href="mailto:krudolph@illinois.edu">w-heller@illinois.edu</a>, or Dr. Sepideh Sadaghiani at (217)300-2566 or <a href="mailto:sepideh@illinois.edu">sepideh@illinois.edu</a>.

If you feel you have not been treated according to the descriptions in this form, or if you have any questions about your rights as a research subject, including questions, concerns, complaints, or to offer input, you may call the Office for the Protection of Research Subjects (OPRS) at 217-333-2670 or e-mail OPRS at irb@illinois.edu.

# **Agreement:**

By signing this document, I am stating that the nature of the study has been explained to me. I am also stating that I have had the opportunity to ask questions concerning any and all aspects of the procedures involved. I understand that I must be 18 or older to provide consent for my child to participate in this study. I am also aware that participation is voluntary, that I may withdraw my consent at any time, and that if I decide not to have my child participate or decide to withdraw my child's participation, I will not be penalized in any way.

| | 0 | • | • | 1 1 | 1 3 |
|-----------|------------|----|---|-----|-----|
| Name of p | participan | t: | | | |
| Name of p | parent: | | | | |
| Signature | of parent: | | | | |
| Date: | | | | | |

I, the undersigned, hereby consent to have my child be a participant in the project described above.